CLINICAL TRIAL: NCT02380833
Title: The Effectiveness of a Paleolithic Based Diet Compared to MyPlate Guidelines, With and Without Exercise, on Physical Conditioning in Women: a Randomized Controlled Trial.
Brief Title: Effectiveness of a Paleolithic Based Diet Compared to MyPlate Guidelines, With and Without Exercise, in Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clemson University (Other)
Responsible Party: Principal Investigator, Elliot D. Jesch, Assistant Professor, Clemson University
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: IRB2014-457
Record Dates: First submitted 2015-02-16; First posted 2015-03-05 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise; Diet, Paleolithic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MyPlate (Active Comparator): To consume a weight maintenance diet based on the United States Department of Agriculture MyPlate nutrition recommendations for eight weeks.
  Interventions: Behavioral: MyPlate
- MyPlate + Exercise (Active Comparator): To consume a weight maintenance diet based on the United States Department of Agriculture MyPlate nutrition recommendations and aerobic and resistance training four days per week for eight weeks.
  Interventions: Behavioral: MyPlate + Exercise
- Paleolithic (Active Comparator): To consume a weight maintenance diet based on alternative (Paleolithic based) nutrition recommendations for eight weeks.
  Interventions: Behavioral: Paleolithic
- Paleolithic + Exercise (Active Comparator): To consume a weight maintenance diet based on alternative (Paleolithic based) nutrition recommendations and aerobic and resistance training four days per week for eight weeks.
  Interventions: Behavioral: Paleolithic + Exercise

INTERVENTIONS:
Behavioral: MyPlate — To consume a weight maintenance diet based on the United States Department of Agriculture MyPlate nutrition recommendations for eight weeks.
  Arms: MyPlate
Behavioral: MyPlate + Exercise — To consume a weight maintenance diet based on the United States Department of Agriculture MyPlate nutrition recommendations and aerobic and resistance training four days per week for eight weeks.
  Arms: MyPlate + Exercise
Behavioral: Paleolithic — To consume a weight maintenance diet based on alternative (Paleolithic based) nutrition recommendations for eight weeks.
  Arms: Paleolithic
Behavioral: Paleolithic + Exercise — To consume a weight maintenance diet based on alternative (Paleolithic based) nutrition recommendations and aerobic and resistance training four days per week for eight weeks.
  Arms: Paleolithic + Exercise

SUMMARY:
The purpose of this study is to determine the effectiveness of recommending either a Paleolithic based diet or the United States Department of Agriculture MyPlate guidelines with or without exercise on physical conditioning, hormones related to energy metabolism, body composition, resting energy expenditure, blood biomarkers, and urine in young, adult females.

ELIGIBILITY:
Inclusion Criteria:

* body fat percent between 20 and 38
* less than 150 minutes of exercise per week at 4.5 or greater Metabolic Equivalent of Task
* not pregnant, trying to become pregnant or lactating
* non-smoker
* no previous resistance training
* have not been on a diet in the past three months
* no dietary restrictions (food allergies, disease conditions, etc)
* have not lost more than 10 lbs. in the past three months

Exclusion Criteria:

* taking any medication
* women who have had a left breast mastectomy
* do not meet criteria of PAR-Q

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in aerobic conditioning | Baseline and 8 weeks
  Peak oxygen consumption
Change in anaerobic power | Baseline and 8 weeks
  Wingate anaerobic threshold
Change in strength | Baseline and 8 weeks
  Chest press and leg press estimated one repetition maximum

SECONDARY OUTCOMES:
Change in resting energy expenditure | Baseline and 8 weeks
  24 hour kcal and respiratory quotient
Change in urine | Baseline and 8 weeks
  Osmolality
Change in insulin (plasma) | Baseline and 8 weeks
  Radioimmunoprecipitation assay
Change in glucagon (plasma) | Baseline and 8 weeks
  Radioimmunoprecipitation assay
Change in ghrelin (plasma) | Baseline and 8 weeks
  Total and active ghrelin; Radioimmunoprecipitation assay
Change in peptide YY 3-36 (plasma) | Baseline and 8 weeks
  Radioimmunoprecipitation assay
Change in adiponectin (plasma) | Baseline and 8 weeks
  Radioimmunoprecipitation assay
Change in leptin (plasma) | Baseline and 8 weeks
  Radioimmunoprecipitation assay
Change in tumor necrosis factor alpha (plasma) | Baseline and 8 weeks
  ELISA
Change in interleukin 6 (plasma) | Baseline and 8 weeks
  ELISA
Change in undercarboxylated osteocalcin (plasma) | Baseline and 8 weeks
  enzymeimmunoassay
Change in total cholesterol (plasma) | Baseline and 8 weeks
  Colorimetric enzyme assay
Change in HDL cholesterol (plasma) | Baseline and 8 weeks
  Colorimetric enzyme assay
Change in non-HDL cholesterol (plasma) | Baseline and 8 weeks
  Calculated from triacylglycerol, total cholesterol and HDL cholesterol
Change in triacylglycerol (plasma) | Baseline and 8 weeks
  Colorimetric enzyme assay
Change in non-esterified fatty acids (plasma) | Baseline and weeks
  Colorimetric enzyme assay
Change in glucose (plasma) | Baseline and 8 weeks
  Colorimetric enzyme assay
Change in ketones (plasma) | Baseline and 8 weeks
  Colorimetric enzyme assay
Change in fat mass | Baseline and 8 weeks
  Dual energy x-ray absorptiometry
Change in fat free mass | Baseline and 8 weeks
  Dual energy x-ray absorptiometry
Change in bone mass | Baseline and 8 weeks
  Dual energy x-ray absorptiometry

OTHER OUTCOMES:
Change in free living activity | Baseline and 8 weeks
  Armband activity monitor worn on the upper left arm (METs)
Change in blood pressure | Baseline and 8 weeks
  Systolic and diastolic blood pressure
Change in resting heart rate | Baseline and 8 weeks
  Beats per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Clemson University, Clemson, South Carolina, United States